CLINICAL TRIAL: NCT04382573
Title: CDK13 Related Disorder : Clinical Phenotype, Neuropsychological Profile, Brain MRI Characteristics and Epigenetic Signature.
Brief Title: Better Delineation of CDK13 Related Phenotype and Epigenetic Signature.
Acronym: CDK13
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0279
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Congenital Heart Defects; Dysmorphic Facial Features and Intellectual Developmental Disorder
Keywords: CDK13-related disorder
MeSH Terms: conditions — Heart Defects, Congenital; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CDK13: CDK13 intragenic pathogenic variant
  Interventions: Genetic: Epigenetic signatures

INTERVENTIONS:
Genetic: Epigenetic signatures — Epigenetic signatures (Dr Sadikovic' lab, London, Ontario, Canada)

SUMMARY:
CDK13 related disorder is mainly characterised by developmental delay (DD) and intellectual disability (ID), ranging from mild to severe, and malformation syndrome.

The aims of this study are first to better delineate the clinical phenotype, as well as the neuropsychological profile, and the brain MRI characteristics; and, second, to study the epigenetic signatures in a cohort of individuals with CDK13 intragenic pathogenic variants. This work will conduct to a MD thesis of a clinical resident geneticist in France.

Physician that will participate will fill an Excel sheet regarding the clinical and neuropsychological assessment.

The investigators will be also happy to have either CD-ROM or a link to have access to the brain MRI data as well as a DNA sample with a minimum 0.5ug of peripheral blood genomic DNA. The investigators will gather the DNA in Montpellier genetic lab (Dr Mouna BARAT) and send the batch to the Dr Sadikovic' lab.

Between 2019 and 2020, The investigators have already recruited data from individuals with CDK13 pathogenic variants from France and several European genetic centres.

DETAILED DESCRIPTION:
The investigators aim to better understand and delineate the genetic syndrome CDK13 This genetic disorder was described in Sepember 2016 in Nature Genetics (PMID 27479907).

Since this first publication of 6 individuals carrying the pathogenic mutation CDK13, 37 other individuals carrying a pathogenic mutation of CDK13 have been reported in the litterature The investigators are seeking to better define the phenotype of individuals with pathogenic variants of CDK13, to better understand intellectual functioning as well as the strengths and weaknesses of intellectual functioning by collecting standardized neuropsychological assessments already performed such as WPPSI/WISC and WAIS. For this purpose, The investigators will gather clinical and neuropsychological data already carried out in the context of care.

The investigators also aim to gather the cerebral MRI scans already performed in order to better delimit the cerebral anomalies observed in individuals and if the sequence is adapted, The investigators will perform VBM studies.

Finally, The investigators will attempt to identify an epigenetic signature in this genetic disease. To this end, The investigators will collect genomic DNA from peripheral blood already collected for genetic analysis and send an anonymized batch of samples to our collaborator, Dr. Bekim Sadicovik. Dr. Bekim Sadicovik and his team will compare the epigenetic DNA methylation-type markers with the corresponding sex and age controls. If specific probes are abnormally methylated in CDK13 individuals, this will determine a disease-specific epigenetic signature. The investigators will then be able to propose an epigenetic signature for individuals with uncharacterized CDK13 variations (class 3, VUS). This method will make it possible to define whether the variation is responsible for the disease or not without going through functional analysis steps that are difficult to implement routinely.

The expected benefits are a better understanding of CDK13 disease, keys to neuropsychological rehabilitation, a better understanding of human brain functions, the possibility of proposing an epigenetic signature for people in whom it is not possible to decide whether a variation in the CDK13 gene is pathological or not

ELIGIBILITY:
Inclusion criteria:

- CDK13 intragenic pathogenic SNV (Single Nucleotide Variant)

Exclusion criteria:

* no pathogenic SNV in CDK13
* no consent for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with CDK13 intragenic pathogenic SNV (Single Nucleotide Variant)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of clinical data | 1 day
  Clinical data such as growth parameters, facial, neurological, ENT, eye, cardiac, etc.. features
Neuropsychological test | 1 day
  Neuropsychological test with total IQ and subscore data using WISC or WAIS test

SECONDARY OUTCOMES:
Evolution of genetic data | 1 day
  Evolution of genetic data : Epigenetic signatures

CONTACTS AND LOCATIONS:
Overall Officials: David GENEVIEVE, Principal Investigator — Department of Medical Genetics
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC